CLINICAL TRIAL: NCT00928759
Title: Etiological Factors of Obesity-Associated Hyperandrogenemia in Peripubertal Girls
Acronym: CRM002
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Other Study IDs: 13552; P50HD028934 (NIH)
Record Dates: First submitted 2008-10-28; First posted 2009-06-26 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Hyperandrogenemia; Polycystic Ovary Syndrome
Keywords: Obesity; Polycystic Ovary Syndrome
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- peripubertal obese girls: Peripubertal obese girls, aged 8 - 16 years, who are obese (BMI-for-age percentile greater or equal to 95)

SUMMARY:
The purpose of this study is to learn if obese pre- and early pubertal girls with hyperandrogenemia (HA) are more insulin resistant (i.e., have lower insulin-stimulated glucose disposal) compared to obese peripubertal girls without HA; and that overnight mean luteinizing hormone (LH) concentration is also an independent predictor of free testosterone concentrations, especially in mid- to late pubertal girls.

DETAILED DESCRIPTION:
A number of pathophysiological mechanisms underlie the polycystic ovary syndrome (PCOS). Neuroendocrine abnormalities play a significant role in most women with PCOS, and PCOS is associated with relative resistance of the gonadotropin releasing hormone (GnRH) pulse generator to negative feedback by progesterone and estradiol. This hypothalamic resistance to negative feedback appears to be a result of hyperandrogenemia (HA), and can also occur in adolescents with HA. We have hypothesized that peripubertal HA (which can represent a forerunner of adult PCOS) can promote the development of PCOS in part via induction of hypothalamic resistance to negative feedback. However, the cause of peripubertal HA remains largely unknown. Obesity is a well-recognized pathophysiological factor in the HA of adult PCOS; and recent data demonstrate that peripubertal obesity is associated with HA. However, the mechanisms underlying the relationship between peripubertal obesity and HA-and the marked variability of androgen levels observed among obese girls-are unknown. We have gathered preliminary data that suggests that obese pre- and early pubertal girls with high androgen levels also exhibit greater degrees of insulin resistance compared to obese girls with lower androgens.

The primary goal of this pilot project is to begin to establish the relationship between insulin resistance (as determined by insulin clamp studies) and free testosterone concentrations in obese peripubertal girls. Secondarily, the aim is to assess the contributions of elevated luteinizing hormone (determined by frequent blood sampling for LH) in obesity-associated HA across puberty.

Subjects will be admitted to the General Clinical Research Center at 1600 h after 4 hours of fasting. We will measure luteinizing hormone every 10 minutes from 1800 h to 0900 h; other hormones (e.g., testosterone) will be assessed as well. Measurements of insulin and glucose will occur before and after a standardized mixed meal (eaten at 1900 h) and while fasting the following morning. A standard hyperinsulinemic euglycemic clamp procedure will be performed from 0900-1100 h.

Characterization of the factors underlying peripubertal HA may permit prediction of which pre- and early pubertal girls will subsequently go on to develop symptoms of PCOS. Data generated by this project will prompt novel future studies to investigate the complex interactions among metabolic and classical endocrine pathways that lead to PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Peripubertal (Tanner stage 1 to 5) girl, age 8-16 years
* Obesity (BMI-for-age ≥ 95th percentile)
* Generally healthy (save for exogenous obesity)
* Ability and willingness of subject/parents to provide informed assent/consent

Exclusion Criteria:

* Age < 8 or > 16 y
* Greater than 4 y post-menarche
* Obesity associated with a diagnosed (genetic) syndrome (e.g., Prader-Willi syndrome, leptin deficiency), obesity related to medications (e.g., glucocorticoids), etc.
* Pregnancy or lactation
* Virilization
* Total testosterone > 150 ng/dl, which suggests the possibility of a virilizing neoplasm
* DHEAS greater than twice upper limit of age-appropriate normal range
* 17-OHP greater than 250 ng/dl, which suggests the possibility of congenital adrenal hyperplasia (if postmenarcheal, the 17-OHP will be collected during the follicular phase, or > 60 if oligomenorrheic) NOTE: If a 17-OHP > 250 ng/dl is confirmed on repeat testing, an ACTH stimulation test will be offered, with a post-ACTH 17-OHP < 1000 ng/dl being required for study participation
* History of premature adrenarche (i.e., appearance of pubic and/or axillary hair before age 8)
* Fasting glucose > 125 mg/dl or hemoglobin A1c > 7.0%
* Abnormal TSH or prolactin
* Evidence of Cushing's syndrome by history or physical exam (e.g., history of impaired growth, striae)
* Hematocrit < 36% or hemoglobin < 12 g/dl
* Significant and current cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring systemic intermittent corticosteroids; etc.)
* Abnormal liver enzymes, age-specific alkaline phosphatase, or a bilirubin > 1.5 times upper limit of normal
* Abnormal sodium, potassium, bicarbonate concentrations, or elevated creatinine concentration
* Weight less than 34 kg is an exclusion criterion (to ensure safe blood withdrawal)
* Subjects using restricted medication (see restrictions below) are excluded unless the subject's primary care provider approves stopping the medication

Ages: 8 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Generally healthy peripubertal girls ages 8 - 16 years with a BMI of > or = to 95th percentile will be recruited from the general population of the surrounding area.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Morning free testosterone | 0700 to 0900 hours
Insulin-stimulated glucose disposal | 0900 to 1100 hours

SECONDARY OUTCOMES:
Estimated 24-hour mean insulin concentration | 24 hours
Luteinizing hormone pulse frequency | 1800 to 0900 hours
Mean luteinizing hormone concentration | 1800 to 0900 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD

REFERENCES:
- [Derived] Burt Solorzano CM, Knudsen KL, Anderson AD, Hutchens EG, Collins JS, Patrie JT, Marshall JC, McCartney CR. Insulin Resistance, Hyperinsulinemia, and LH: Relative Roles in Peripubertal Obesity-Associated Hyperandrogenemia. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2571-2582. doi: 10.1210/jc.2018-00131. PMID 29897474